CLINICAL TRIAL: NCT01517009
Title: A Multicenter Phase II Study of Neoadjuvant Docetaxel, Cisplatin and Capecitabine and Protocolized Surgery in Resectable Gastric Cancer
Acronym: DoCCS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jeroen Bosch Ziekenhuis (Other)
Collaborators: Eindhoven Cancer Registry (Other)
Responsible Party: Principal Investigator, Anneriet Dassen, Ms A.E. Dassen, MD, Principle Investigator, Jeroen Bosch Ziekenhuis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DoCCS; Dutch trialregister (Registry Identifier: NTR2306); 2007-007273-23 (EudraCT Number)
Record Dates: First submitted 2011-10-21; First posted 2012-01-25 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Gastric Cancer
Keywords: Neo-adjuvant chemotherapy; D1extra-resection
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Docetaxel — 60 mg/m2, 1 gift every 3 weeks, in total 4 gifts
  Other Names: Taxotere
Drug: cisplatin — 60 mg/m2, one gift every three weeks, in total 4 gift
Drug: Capecitabine — 1875 mg/m2 in two equally divided doses day 1-14, repeated every three weeks, in total 4 cycles
  Other Names: Xeloda
Procedure: D1extra-resection — An extended lymphadenectomy compared to a D1 resection for gastric cancer

SUMMARY:
The purpose of this study is to determine the feasibility of chemotherapy, consisting of docetaxel, cisplatin and capecitabine given prior to surgery for stomach cancer. Furthermore, an extended type of removal of lymph nodes will be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Ib-IVa histological proven resectable gastric adenocarcinoma, including gastro-oesophageal junction/cardia carcinoma Siewert 2 and 3
* ASA 2 or less
* Age 18 years or more
* No prior radio- or chemotherapy conflicting with the treatment of gastric cancer
* Haematology/Renal function/Liver function within designated range
* Patient's consent form obtained, signed and dated before beginning specific protocol procedures
* absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* before patient registration/randomization, written informed consent must be given according to GCP, WMO and local regulations.

Exclusion Criteria:

* Previous or other current malignancies, with the exception of adequately treated in situ carcinoma of the cervix uteri or non-melanoma skin cancer
* Other current serious illness or medical conditions
* Severe cardiac illness (NYHA class III-IV)
* Significant neurologic or psychiatric disorders
* Uncontrolled infections
* Active DIC
* Other serious underlying medical conditions that could impair the ability of the patient to participate in the study
* Known hypersensitivity to docetaxel (or any drug formulated with Polysorbate-80), or cisplatin or capecitabine or 5-FU
* Definite contraindications for the use of corticosteroids
* Use of immunosuppressive or antiviral drugs
* Any other experimental drugs within a 4-week period prior to start of neoadjuvant chemotherapy and throughout the study period
* Pregnant or lactating women
* Patients with reproductive potential not implementing adequate contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-06; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The number of patients with (serious) adverse events receiving the combination of 4 courses of docetaxel, cisplatin and capecitabine as neoadjuvant chemotherapy and standardized surgery in resectable localized or locally advanced gastric cancer. | 18 weeks
  Patients receive every 3 weeks a cycle of chemotherapy, in total 4 cylcles will be given. Surgery will be performed approximately 6 weeks after the last cycle.

SECONDARY OUTCOMES:
The number of patients receiving a D1-extra-resection as protocolized surgery in resectable gastric cancer | 30 days

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - VieCuri Hospital, Venlo, Limburg
  - Jeroen Bosch Hospital, 's-Hertogenbosch, North Brabant
  - Catharina Hospital, Eindhoven, North Brabant
  - Elkerliek Hospital, Helmond, North Brabant
  - Maxima Medical Centre, Veldhoven, North Brabant